CLINICAL TRIAL: NCT01311895
Title: Randomized Clinical Trial Comparing Two Protocols Using IV Hydromorphone
Brief Title: Clinical Trial Comparing Two Protocols Using Intravenous (IV) Hydromorphone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMC 10-07-201
Record Dates: First submitted 2011-03-04; First posted 2011-03-10 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Acute Pain
Keywords: acute; pain; emergency department; hydromorphone
MeSH Terms: conditions — Acute Pain; Pain; Emergencies | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- H2O (Experimental): 2 mg IV hydromorphone administered over 2-3 minutes as initial dose
  Interventions: Drug: H2O
- 1+1 (Experimental): 1 mg IV hydromorphone followed by an additional 1 mg IV hydromorphone 15 minutes later if the patient answers "yes" to the following question: "Do you want more pain medication?"
  Interventions: Drug: 1+1

INTERVENTIONS:
Drug: H2O — 2 mg IV hydromorphone
  Other Names: Dilaudid
  Arms: H2O
Drug: 1+1 — 1mg I hydromorphone followed by an optional 1 mg IV hydromorphone 15 minutes later if the patient answers "yes" to the question, "Do you want more pain medication?"
  Other Names: Dilaudid
  Arms: 1+1

SUMMARY:
The purpose of this study is to compare two opioid protocols ("H2O" and "1+1") for the treatment of acute severe pain in the emergency department. The investigators primary hypothesis is that the "H2O" protocol will be more efficacious than the "1+1" protocol in Emergency Department patients aged 21-64 years. The primary outcome is the proportion of patients in each arm who choose to forgo additional pain medication at 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 21 years and less than 65 years: This is a study of non-elderly adult patients. In addition, patients aged 21 years and younger are automatically triaged to the Children's Emergency Department (ED).
2. Pain with onset within 7 days: Pain within seven days is the definition of acute pain that has been used in ED literature.
3. ED attending physician's judgment that patient's pain warrants intravenous (IV) opioids

Exclusion Criteria:

1. Use of other opioids or tramadol within past 24 hours: to avoid introducing assembly bias related to recent opioid use, since this may affect baseline levels of pain and need for analgesics.
2. Prior adverse reaction to opioids.
3. Chronic pain syndrome: frequently recurrent or daily pain for at least 3 months results in modulation of pain perception which is thought to be due to down-regulation of pain receptors. Examples of chronic pain syndromes include sickle cell anemia, osteoarthritis, fibromyalgia, and peripheral neuropathies.
4. Alcohol intoxication: the presence of alcohol intoxication as judged by the treating physician may alter pain perception.
5. Systolic Blood Pressure <90 mm Hg: Opioids can produce peripheral vasodilation that may result in orthostatic hypotension.
6. Oxygen saturation < 95% on room air: For this study, oxygen saturation must be 95% or above on room air in order to be enrolled.
7. Use of monoamine oxidase (MAO) inhibitors in past 30 days: MAO inhibitors have been reported to intensify the effects of at least one opioid drug causing anxiety, confusion and significant respiratory depression or coma.
8. CO2 measurement greater than 46: In accordance with standard protocol, three subsets of patients will have their CO2 measured using a handheld capnometer prior to enrollment in the study. If the CO2 measurement is greater than 46 then the patient will be excluded from the study. The 3 subsets are as follows:

   * All patients who have a history of chronic obstructive pulmonary disease (COPD)
   * All patients who report a history of asthma together with greater than a 20 pack-year smoking history
   * All patients reporting less than a 20 pack-year smoking history who are having an asthma exacerbation

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center Moses Division Emergency Department, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- H2O (2 mg IV Hydromorphone): 2 mg IV hydromorphone
  H2O: 2 mg intravenous (IV) hydromorphone
- 1+1 (1 mg IV Hydromorphone + Optional 1 mg IV Hydromorphone): 1 mg intravenous (IV) hydromorphone followed by an additional 1 mg IV hydromorphone 15 minutes later if the patient answers "yes" to the following question: "Do you want more pain medication?"
  1+1: 1mg I hydromorphone followed by an optional 1 mg IV hydromorphone 15 minutes later if the patient answers "yes" to the question, "Do you want more pain medication?"
Period: Overall Study
Arm/Group | H2O (2 mg IV Hydromorphone) | 1+1 (1 mg IV Hydromorphone + Optional 1 mg IV Hydromorphone)
Started | 175 | 175
Completed | 175 | 175
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The discrepancy between the number of patients enrolled and randomized and those included in analysis is due to the following.
  H2O group: never given IV opioids (2), received ketorolac or additional opioids within the 60 min (7).
  1+1 group: missing data (3), didn't receive 2nd dose within 60 min (2), received additional opioids within 60 min (2)
Groups:
- H2O (2 mg IV Hydromorphone): 2 mg IV hydromorphone
  H2O: 2 mg IV hydromorphone
- 1+1 (1 mg IV Hydromorphone + Optional 1 mg IV Hydromorphone): 1 mg IV hydromorphone followed by an additional 1 mg IV hydromorphone 15 minutes later if the patient answers "yes" to the following question: "Do you want more pain medication?"
  1+1: 1mg I hydromorphone followed by an optional 1 mg IV hydromorphone 15 minutes later if the patient answers "yes" to the question, "Do you want more pain medication?"
- Total: Total of all reporting groups
Arm/Group | H2O (2 mg IV Hydromorphone) | 1+1 (1 mg IV Hydromorphone + Optional 1 mg IV Hydromorphone) | Total
Number analyzed (Participants) | 166 | 168 | 334
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [33 to 52] | 42 [33 to 50] | 43 [33 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 107 | 210
  Male | 63 | 61 | 124
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 109 | 116 | 225
  Black | 48 | 44 | 92
  White | 8 | 5 | 13
  Other | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 166 | 168 | 334
Weight [Median (Inter-Quartile Range); unit: lbs] | 180 [165 to 210] | 186 [170 to 219] | 184 [165 to 219]
Location of pain [Count of Participants; unit: Participants]
  Abdomen | 116 | 112 | 228
  Other | 50 | 56 | 106
Pain intensity [Count of Participants; unit: Participants] — Pain intensity is measured on the numerical rating scale (NRS) from 0 ("no pain") to 10 ("worst pain imaginable").
  Participants
    3-7 | 28 | 26 | 54
    8 | 24 | 28 | 52
    9 | 16 | 22 | 38
    10 | 98 | 92 | 190
Nauseated or vomited before receiving opioids in the Emergency Department (ED) [Count of Participants; unit: Participants]
  Yes | 108 | 105 | 213
  No | 58 | 63 | 121

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Satisfactory Pain Management at 60 Minutes
Description: The primary outcome is the proportion of patients in each arm who choose to forgo additional pain medication at 60 minutes. This is defined as the number of patients who declined additional pain medication at 60 minutes.
Time Frame: 60 minutes
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- H2O (2 mg IV Hydromorphone): 2 mg IV hydromorphone administered over 2-3 minutes as initial dose
  H2O: 2 mg IV hydromorphone
Arm/Group | H2O (2 mg IV Hydromorphone) | 1+1 (1 mg IV Hydromorphone + Optional 1 mg IV Hydromorphone)
Number analyzed (Participants) | 166 | 168
Participants | 112 | 113

2. Secondary Outcome: Mean Change in Pain Intensity From Baseline to 60 Minutes
Description: Pain intensity is measured in numerical rating scale (NRS) units from 0 ("no pain") to 10 ("worst pain imaginable"). The change here represents the NRS score given by the patients at 60 minutes subtracted from the score at baseline, before treatment in the Emergency Department.
Time Frame: 60 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | H2O (2 mg IV Hydromorphone) | 1+1 (1 mg IV Hydromorphone + Optional 1 mg IV Hydromorphone)
Number analyzed (Participants) | 166 | 168
units on a scale | 6.1 (3.1) | 5.7 (3.0)

3. Secondary Outcome: Number of Patients Who Reported no Pain or Mild Pain at 60 Minutes
Time Frame: 60 minutes
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | H2O (2 mg IV Hydromorphone) | 1+1 (1 mg IV Hydromorphone + Optional 1 mg IV Hydromorphone)
Number analyzed (Participants) | 166 | 168
Participants | 112 | 112

ADVERSE EVENTS:
Time Frame: 60 minutes
Description: The discrepancy between the number of patients enrolled and randomized and those included in analysis is due to the following.
  H2O group: never given IV opioids (2), received ketorolac or additional opioids within the 60 min (7).
  1+1 group: missing data (3), didn't receive 2nd dose within 60 min (2), received additional opioids within 60 min (2)
Arm/Group | H2O (2 mg IV Hydromorphone) | 1+1 (1 mg IV Hydromorphone + Optional 1 mg IV Hydromorphone)
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/168
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/168
Other Adverse Events (participants affected / at risk) | 56/166 | 53/168
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | H2O (2 mg IV Hydromorphone) (N=166) | 1+1 (1 mg IV Hydromorphone + Optional 1 mg IV Hydromorphone) (N=168)
Administration of naloxone (Endocrine disorders) | 0 | 0
Oxygen saturation <95% (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulse rate <50 beats/min (Cardiac disorders) | 0 | 5
Systolic blood pressure <90 mmHg (Vascular disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 28 | 20
Nausea (Gastrointestinal disorders) | 17/58 | 17/63 — excludes patients who were nauseated or vomiting before receiving opioids
Vomiting (Gastrointestinal disorders) | 9/58 | 8/63 — excludes patients who were nauseated or vomiting before receiving opioids in the ED

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes